CLINICAL TRIAL: NCT04595682
Title: Estradiol Effects on Behavioral and Reward Sensitivity to Alcohol Across the Menstrual Cycle
Brief Title: Estradiol Effects on Alcohol Across the Menstrual Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Fillmore (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Mark Fillmore, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 52637; 1R01AA027990-01A1 (NIH)
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use, Unspecified
Keywords: estradiol; reward; menstrual; hormone
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- menstrual cycle (Experimental): Participants will have their alcohol sensitivity test once during their early follicular phase and once during their late follicular phase
  Interventions: Drug: Placebo; Drug: Alcohol

INTERVENTIONS:
Drug: Placebo — Participants will attend two identical laboratory sessions to test sensitivity to the rewarding and disinhibiting effects of a controlled dose of alcohol, once during the early follicular phase and once during the late follicular phase. The test battery consists of measures of rewarding effects and alcohol (or placebo) effects on disinhibition and impulsive choice. The placebo consists of 300 ml of lemon-flavored soda with a small amount (3 ml) of alcohol floated on top.
Drug: Alcohol — Participants will attend two identical laboratory sessions to test sensitivity to the rewarding and disinhibiting effects of a controlled dose of alcohol, once during the early follicular phase and once during the late follicular phase. The test battery consists of measures of rewarding effects and alcohol effects on disinhibition and impulsive choice. The alcohol dose consists of 0.60 g/kg absolute alcohol that produces a peak blood-alcohol concentration of 80 mg/dl. Doses will be mixed with a carbonated, non-caffeinated, lemon-flavored soda and consumed within 10 minutes.

SUMMARY:
This study will provide the first rigorous integrative test of the hypothesis that rapid rises in estradiol (a female hormone) increase the rewarding and disinhibiting effects of alcohol and that such increased sensitivity correlates with increased alcohol use. Identification of the behavioral mechanisms by which estradiol surges can increase alcohol use would provide a critical advancement of neurobiological theory of alcohol abuse in women, an understudied area, as well as provide new directions for personalization of alcohol abuse treatment in women.

In this study, naturally-cycling women will be examined daily over their menstrual cycle using an integrative combination of daily ecological assessments of hormone fluctuations and alcohol use along with strategically-timed laboratory tests of their acute sensitivity to the rewarding and disinhibiting effects of a controlled dose of alcohol.

DETAILED DESCRIPTION:
A longitudinal study design will test hormonal influences across the menstrual cycle on women's naturalistic drinking behavior, as well as their acute sensitivity to the rewarding and disinhibiting effects of alcohol in the laboratory, two key mechanisms of its abuse potential. Subjects will attend a diagnostic visit to assess baseline clinical characteristics. In addition, subjects will attend two laboratory visits to test alcohol sensitivity at two key points in the cycle: during the early follicular phase when E2 is low and the late follicular phase when E2 is rising (see Figure 6). Every day after their first laboratory visit for 35 consecutive days, women will provide saliva samples each morning to assess hormonal levels and complete a self-report on their drinking behavior and alcohol craving every evening through a secure online server. The daily saliva and self-report data will allow fine-grained investigation of the lagged correlations between E2 and daily alcohol use patterns and alcohol craving across the menstrual cycle. The two laboratory visits will test and compare the acute sensitivity to rewarding and disinhibiting effects of a controlled dose of alcohol during the early follicular phase when E2 is low and the late follicular phase when E2 is rising. Volunteers will be followed daily to assess when they start their next menstrual cycle (i.e., the day they start bleeding). Within 1-2 days of that point, volunteers are scheduled to attend their initial diagnostic visit. Participants are then counterbalanced to begin the study during either their early follicular phase (approximately day 5) or their late follicular phase (approximately day 12) which is also when they begin their 35 days of consecutive daily data collection. This serves to counterbalance the order of the two alcohol sensitivity test sessions: early follicular versus late follicular phase. Ovulation testing and daily salivary E2 will confirm the proximity of the late follicular phase to ovulation, with the goal of ovulation occurring 1-3 days after the late follicular visit, and capturing a higher, rising E2 level in the late follicular phase relative to a lower level in the early follicular phase.

ELIGIBILITY:
Inclusion Criteria:

* female
* regular menstrual cycle
* consume alcohol at least once per week
* no history of drug or alcohol dependence

Exclusion Criteria:

* use of hormone-based medications
* irregular menstrual cycle
* current pregnancy
* primary sensorimotor handicap
* frank neurological disorder
* pervasive developmental disorder
* frank psychosis
* diagnosed intellectual disability
* medical condition contraindicating alcohol use
* substance abuse history (except nicotine)
* body mass index (BMI) 30 or above
* alcohol abstainer

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fillmore, PhD, Principal Investigator — University of Kentucky; Michelle Martel, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University Of Kentucky Psychology Research Lab, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griffith AK, Martel MM, Fillmore MT. Effect of menstrual cycle on rewarding properties of alcohol cues in women. Psychol Addict Behav. 2024 Sep;38(6):676-687. doi: 10.1037/adb0000978. Epub 2023 Dec 7. PMID 38059946
- [Derived] Griffith AK, Martel MM, Eisenlohr-Moul T, Fillmore MT. Heightened sensitivity to the disinhibiting effect of alcohol in women during the late follicular phase of the menstrual cycle. Exp Clin Psychopharmacol. 2023 Aug;31(4):839-848. doi: 10.1037/pha0000611. Epub 2022 Oct 20. PMID 36265052

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For this study participants are randomly started in Late Follicular Phase (Day 12) or Early Follicular Phase (Day 5) based on when they are enrolled in the study and which day of their menstrual cycle they are on when enrolled. This order does not affect the treatment given to each participant in any way. Every participant is given a placebo, then alcohol.
Groups:
- Late Follicular Phase Visit First, Then Early Follicular Phase Visit: Participants in this group will track their menstrual cycle, provide daily saliva samples, and undergo two rounds of alcohol sensitivity testing (with both placebo and alcohol).
  beginning the study during their late follicular phase (approximately day 12) which is also when they begin their 35 days of consecutive daily data collection
- Early Follicular Phase Visit First, Then Late Follicular Phase Visit: Participants in this group will track their menstrual cycle, provide daily saliva samples, and undergo two rounds of alcohol sensitivity testing (with both placebo and alcohol).
  beginning the study during their early follicular phase (approximately day 5) which is also when they begin their 35 days of consecutive daily data collection
Period: Overall Study
Arm/Group | Late Follicular Phase Visit First, Then Early Follicular Phase Visit | Early Follicular Phase Visit First, Then Late Follicular Phase Visit
Started | 45 | 55
Completed | 45 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Participants in this group will track their menstrual cycle, provide daily saliva samples, and undergo two rounds of alcohol sensitivity testing (with both placebo and alcohol).
Arm/Group | Study Participants
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.98 (3.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 80
  More than one race | 10
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Attentional Bias (Early Follicular Phase)
Description: Attentional bias is measured by the visual dot-probe task and provides an implicit assessment of the rewarding properties of alcohol as indicated by the degree to which an acute dose of alcohol increases the drinker's attention to alcohol cues is measured. Subjects look at images on a screen and their attention to various images is measured. An alcohol-related image and a neutral control image are presented briefly side-by-side, on a computer screen. An eye tracker embedded into the monitor provides an unobtrusive measure of the duration (dwell time) that volunteers look at each image.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Study Participants
Number analyzed (Participants) | 100
milliseconds
  Alcohol | 347.99 (51.61)
  Placebo | 355.02 (56.02)

2. Primary Outcome: Attentional Bias (Late Follicular Phase)
Description: as for outcome 1
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Study Participants
Number analyzed (Participants) | 100
milliseconds
  Alcohol | 356.01 (57.58)
  Placebo | 352.81 (57.14)

3. Primary Outcome: Disinhibition (Early Follicular Phase)
Description: Disinhibition wil be measured by the cued go/no-go task, which requires participants to respond quickly to go targets and inhibit responses to no-go targets. Participants complete 250 trials in which they are presented with a cue, followed by a target. A go target is green, and participants are instructed to press a button when presented with a go target. A no-go target is blue, and participants are instructed to do nothing when this appears.
  A go cue predicts a go target with 80% accuracy, whereas a no-go cue predicts a no-go target with 80% accuracy.
  The condition of interest is when a go cue is followed by a no-go target. The proportion reported is the proportion of trials under this condition in which participants press the button (expecting a go target but presented with a no-go target).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: proportion of inhibition failures
Arm/Group | Study Participants
Number analyzed (Participants) | 100
proportion of inhibition failures
  Alcohol | 0.107 (0.12)
  Placebo | 0.04 (0.06)

4. Primary Outcome: Disinhibition (Late Follicular Phase)
Description: as for outcome 3
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: proportion of inhibition failures
Arm/Group | Study Participants
Number analyzed (Participants) | 100
proportion of inhibition failures
  Alcohol | 0.134 (0.13)
  Placebo | 0.045 (0.06)

5. Primary Outcome: Subjective Ratings of the Rewarding Effects of Alcohol (Early Follicular Phase)
Description: a visual analog scale from 0-100, with 0 being not rewarding at all and 100 being very rewarding
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 100
score on a scale
  Alcohol | 56.99 (25.61)
  Placebo | 39.2 (23.26)

6. Primary Outcome: Subjective Ratings of the Rewarding Effects of Alcohol (Late Follicular Phase)
Description: a visual analog scale from 0-100, with 0 being not rewarding at all and 100 being very rewarding
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 100
score on a scale
  Alcohol | 60.17 (22.23)
  Placebo | 39.43 (22.37)

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT04595682/Prot_SAP_ICF_001.pdf